CLINICAL TRIAL: NCT02543931
Title: Phase Ib Randomized, Double-Blind, Placebo-Controlled Study of Meriva in Rheumatoid Arthritis
Brief Title: Curcuma Longa L in Rheumatoid Arthritis
Acronym: CLaRA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: University of Arizona (Other)
Collaborators: Vanderbilt University (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Janet L. Funk, Associate Professor, University of Arizona
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1501627690; R34AT007837 (NIH)
Record Dates: First submitted 2015-08-06; First posted 2015-09-07 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Rheumatoid Arthritis
Keywords: turmeric; curcumin; curcuminoids; arthritis; methotrexate
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Curcumin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): Participants will take 4 placebo capsules twice a day for one month
  Interventions: Drug: placebo
- Meriva, low dose (Experimental): Participants will take 4 Meriva-250mg capsules twice a day for one month
  Interventions: Drug: Meriva
- Meriva, high dose (Experimental): Participants will take 4 Meriva-500mg capsules twice a day for one month
  Interventions: Drug: Meriva

INTERVENTIONS:
Drug: Meriva — Meriva is an enhanced-bioavailability, curcuminoid-enriched turmeric dietary supplement that is sold over the counter in the United States and other countries.
  Other Names: turmeric, enhanced bioavailability
  Arms: Meriva, high dose; Meriva, low dose
Drug: placebo — Placebo capsules containing inert ingredients
  Other Names: inactive capsule
  Arms: Placebo

SUMMARY:
The purpose of this study is to find out whether turmeric dietary supplements that are available over the counter for general use in the United States are safe and useful when taken specifically for the treatment of rheumatoid arthritis (RA) and how the active principles in turmeric are broken down and metabolized by the body in individuals with RA.

DETAILED DESCRIPTION:
A placebo-controlled, double-blind, three-arm Phase Ib clinical trial assessing two doses of a commercially available curcuminoid formulation with enhanced bioavailability vs. placebo in a rheumatoid arthritis (RA) population is proposed. The primary aim of this clinical planning study is to determine the dose-dependent tolerability of an enhanced bioavailability curcuminoid formulation in an RA population, including pharmacokinetic analyses, to inform the design of a future Phase II trial assessing the anti-inflammatory efficacy of curcuminoids in the treatment of RA. Secondarily, estimates of effect size for changes in known biomarkers of inflammation in RA will be determined.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Diagnosis of RA (ACR 2010 criteria)
  * Age > 18 years old
  * Active disease at screening visit as defined by:

    * Disease Activity Score [DAS]-28 (4)-erythrocyte sedimentation rate (ESR) > 3.2, and
    * C reactive protein (CRP) > 1.0 mg/dL or ESR > 20.
  * Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Current treatment with any biologic agent (e.g. tumor necrosis factor (TNF) inhibitors: etanercept , infliximab, adalimumab; interleukin 1(IL-1) inhibitors: anakinra ; lymphocyte directed: abatacept, rituximab; and Janus kinase (JAK) inhibitors: tofacitinib).
* Past biologic use allowed if ended > 3 months prior to randomization (> 12 months for Rituximab)
* History of non-response to biologics.
* Disease-modifying anti-inflammatory agents (DMARDs), including methotrexate, hydroxychloroquine, sulfasalazine, and minocycline, will be allowed if stable for 1 month prior to randomization and unchanged throughout the study.
* Leflunomide, gold compounds, azathioprine, or cyclosporine will be exclusionary if used within the month prior to randomization.
* Oral Corticosteroid use > 10 mg/d prednisolone or equivalent or parenteral corticosteroids of any dose will be exclusionary (1 month prior to randomization until final assessment visit).

  * Oral corticosteroids in low doses (< 10 mg/d prednisone or equivalent) will be allowed if stable for 1 month prior to randomization and unchanged throughout the study).
  * Topical, inhaled, or intranasal steroids are not exclusionary
  * Past parenteral or oral (> 10 mg/d prednisolone equivalent) corticosteroids allowed if not used within one month prior to randomization
* Non-steroidal anti-inflammatory drugs (NSAID) are exclusionary if used continuously or > 3 doses in 7 days.

  o Enrollment will be allowed after a washout period of 1 week prior to randomization for use of >3 doses In 7 days).
* Herbal supplements will be exclusionary.

  o Enrollment will be allowed after a washout period of 1 week prior to randomization). Patients will also be asked to minimize intake of curcuminoid-containing foods during the entire study period.
* History of positive skin test for tuberculosis (TB) without treatment.
* Systemic complications of RA (e.g. vasculitis).
* Recent surgery < 1 month prior, or scheduled surgery < 2 months after randomization
* History of malignancy, other than superficial basal or squamous cell carcinoma of the skin.
* History of, or concurrent, serious chronic infection.
* Women who are pre-menopausal (women with menses within the past 12-months) with an intact uterus must have a negative pregnancy test at screening and randomization, must be using a medically acceptable form of birth control, and may not be breast feeding.
* Worsening or uncontrolled end organ disease or intercurrent illness which, in the opinion of the investigator, may pose an added risk to the patient including, but not limited to, evidence of impaired renal function , hematological, gastrointestinal, endocrine, pulmonary, cardiac, neurologic or psychiatric disease.
* Acute or chronic liver disease, including Gilbert's syndrome.
* History of any atrioventricular (AV) nodal conduction defect or a P-R interval (interval between P wave QRS complex) and on ECG > 0.2 sec.
* Use of illicit drugs or high alcohol consumption or current/recent (within past 5 years) history of drug or alcohol abuse.
* Treatment within 28 days of randomization with another investigational agent,
* Have a history of allergic reactions to turmeric, Meriva, or curcuminoids, including turmeric-containing foods such as curry or mustard.
* Inability or difficulty in swallowing oral medications, or any malabsorption condition.
* Inability to provide informed consent for any reason or to complete simple questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-11; Primary Completion 2017-06 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 1 week and 4 weeks
Area under curve (AUC) | 0-24 h
  Following first dose.
Cmax | 0-24h
  Following first dose.
Tmax | 0-24h
  Following first dose.
T1/2 | 0-24h
  Following first dose.
Cmax | 1 week and 4 week
  Plasma concentration after multiple daily dosings

SECONDARY OUTCOMES:
Changes in biomarkers of inflammation | 1 and 4 weeks
  Changes from baseline in blood levels of ESR and C reactive protein will be determined after 1 and 4 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Janet Funk, MD, Principal Investigator — The University of Arizona
Locations (1):
- The University of Arizona, Tucson, Arizona, United States